CLINICAL TRIAL: NCT00664001
Title: Randomized Double-Blind Placebo-Controlled Trial of Oral Anti-Oxidant Supplementation for the Prevention of Acute Mountain Sickness.
Brief Title: Anti-Oxidant Supplementation for the Prevention of Acute Mountain Sickness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Altitude Physiology Expeditions (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: JK Baillie, Apex
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Anti-oxidant
Record Dates: First submitted 2008-04-07; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Placebo tablet
  Interventions: Dietary Supplement: Matched placebo for anti-oxidant supplementation
- Intervention (Active Comparator): Anti-oxidant supplementation
  Interventions: Dietary Supplement: Anti-oxidant supplementation

INTERVENTIONS:
Dietary Supplement: Anti-oxidant supplementation — Daily dose of 1g L-ascorbic acid, 400 IU of alpha-tocopherol acetate, and 600mg of alpha-lipoic acid in sealed capsules as anti-oxidant supplementation.
  Arms: Intervention
Dietary Supplement: Matched placebo for anti-oxidant supplementation — Matched placebo for anti-oxidant supplementation
  Arms: Control

SUMMARY:
Acute mountain sickness (AMS), high altitude pulmonary edema (HAPE), and high altitude cerebral edema (HACE) are complications of rapid ascent to high altitude. Several features suggest that raised intracranial pressure (ICP) may be an important factor in the pathogenesis of AMS. Magnetic resonance imaging of HACE patients has demonstrated that the oedema in HACE is of the vasogenic, rather that cytotoxic, type. Thus it is likely that cerebrovascular permeability has an important role in the development of AMS and HACE.

Reactive oxygen species (ROS) have been shown to alter the permeability of the blood-brain barrier in severe ischaemia, causing vasogenic cerebral oedema. Endogenous antioxidant systems may have some capacity to respond to oxidative stress in hypoxia. The plasma concentration of urate, a powerful endogenous antioxidant, rises on acute exposure to high altitude and may play a crucial antioxidant role in systemic hypoxia. This antioxidant prevents free-radical induced cerebral oedema in animal models.

There are numerous sources of ROS in hypoxia, including the mitochondrial electron transfer chain, haemoglobin (Hb) autoxidation and xanthine oxidase activity. There have been several reports of raised markers of oxidative stress in humans at moderate altitude (<3000m).

Oral antioxidant supplementation with preparations containing vitamins C and E in humans at altitude has been shown to decrease breath pentanes (a marker of oxidative stress), and improve erythrocyte filterability. In a small randomised controlled trial, Bailey and Davies demonstrated a significant reduction in symptoms of AMS in subjects taking an oral antioxidant cocktail.

The antioxidants alpha-lipoic acid, vitamin C and vitamin E act synergistically to provide membrane protection from free radical damage, and may protect against hypoxia-induced vascular leakage. We hypothesised that this combination of antioxidants would reduce the severity of acute mountain sickness, and reduce pulmonary artery pressures, in healthy lowlanders acutely exposed to high altitude.

DETAILED DESCRIPTION:
Acute mountain sickness (AMS), high altitude pulmonary edema (HAPE), and high altitude cerebral edema (HACE) are complications of rapid ascent to high altitude. By definition, AMS is a benign condition, but it is likely that the same pathology underlies high altitude cerebral oedema (HACE). In contrast, HAPE occurs in the context of pathologically elevated pulmonary artery pressures and uneven distribution of hypoxic pulmonary vasoconstriction across the pulmonary vascular bed.

Several features suggest that raised intracranial pressure (ICP) may be an important factor in the pathogenesis of AMS. Magnetic resonance imaging of HACE patients has demonstrated that the oedema in HACE is of the vasogenic, rather that cytotoxic, type. Thus it is likely that cerebrovascular permeability has an important role in the development of AMS and HACE.

Reactive oxygen species (ROS) have been shown to alter the permeability of the blood-brain barrier in severe ischaemia, causing vasogenic cerebral oedema. Endogenous antioxidant systems may have some capacity to respond to oxidative stress in hypoxia. The plasma concentration of urate, a powerful endogenous antioxidant, rises on acute exposure to high altitude and may play a crucial antioxidant role in systemic hypoxia. This antioxidant prevents free-radical induced cerebral oedema in animal models.

The pathogenesis of HAPE is understood to have two components: (i) increased pulmonary arterial pressures secondary to hypoxic pulmonary vasoconstriction and; (ii) an increase in endothelial permeability, possibly due to stress rupture of pulmonary capillaries. There is much debate surrounding the cellular mechanisms of hypoxic pulmonary vasoconstriction, but it is likely that ROS have an important role.

There are numerous sources of ROS in hypoxia, including the mitochondrial electron transfer chain, haemoglobin (Hb) autoxidation and xanthine oxidase activity. There have been several reports of raised markers of oxidative stress in humans at moderate altitude (<3000m).

Oral antioxidant supplementation with preparations containing vitamins C and E in humans at altitude has been shown to decrease breath pentanes (a marker of oxidative stress), and improve erythrocyte filterability. In a small randomised controlled trial, Bailey and Davies demonstrated a significant reduction in symptoms of AMS in subjects taking an oral antioxidant cocktail.

The antioxidants alpha-lipoic acid, vitamin C and vitamin E act synergistically to provide membrane protection from free radical damage, and may protect against hypoxia-induced vascular leakage. We hypothesised that this combination of antioxidants would reduce the severity of acute mountain sickness, and reduce pulmonary artery pressures, in healthy lowlanders acutely exposed to high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Apex 2 trial

Exclusion Criteria:

* High altitude pulmonary oedema (HAPE)
* Gasto-intestinal illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2003-03; Primary Completion 2003-08 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Acute Mountain Sickness (AMS) as assessed by Lake Louise Consensus symptom score | Day 2

SECONDARY OUTCOMES:
Pulmonary artery systolic pressure | Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Baillie, Principal Investigator — Apex Bioscience
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Hall DP, MacCormick IJ, Phythian-Adams AT, Rzechorzek NM, Hope-Jones D, Cosens S, Jackson S, Bates MG, Collier DJ, Hume DA, Freeman T, Thompson AA, Baillie JK. Network analysis reveals distinct clinical syndromes underlying acute mountain sickness. PLoS One. 2014 Jan 22;9(1):e81229. doi: 10.1371/journal.pone.0081229. eCollection 2014. PMID 24465370
- [Derived] MacCormick IJ, Somner J, Morris DS, MacGillivray TJ, Bourne RR, Huang SS, MacCormick A, Aspinall PA, Baillie JK, Thompson AA, Dhillon B. Retinal vessel tortuosity in response to hypobaric hypoxia. High Alt Med Biol. 2012 Dec;13(4):263-8. doi: 10.1089/ham.2011.1097. PMID 23270443
- [Derived] Baillie JK, Thompson AA, Irving JB, Bates MG, Sutherland AI, Macnee W, Maxwell SR, Webb DJ. Oral antioxidant supplementation does not prevent acute mountain sickness: double blind, randomized placebo-controlled trial. QJM. 2009 May;102(5):341-8. doi: 10.1093/qjmed/hcp026. Epub 2009 Mar 9. PMID 19273551
- See also: Related Info — http://altitude.org